CLINICAL TRIAL: NCT01332656
Title: A Phase 2, Multi-Center, Double-Blind, Placebo Controlled, Randomized Study of Ombrabulin in Patients With Platinum-Sensitive Recurrent Ovarian Cancer Treated With Carboplatin/Paclitaxel
Brief Title: Study of Ombrabulin in Patients With Platinum-Sensitive Recurrent Ovarian Cancer Treated With Carboplatin/Paclitaxel
Acronym: OPSALIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC10260; 2010-024631-16 (EudraCT Number); U1111-1118-5437 (Other: UTN)
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-11

CONDITIONS: Ovarian Cancer Recurrent
MeSH Terms: interventions — AC 7700; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Ombrabulin, Paclitaxel and Carboplatin
  Interventions: Drug: Ombrabulin (AVE8062); Drug: Paclitaxel; Drug: Carboplatin
- Arm B (Placebo Comparator): Placebo, Paclitaxel and Carboplatin
  Interventions: Drug: Placebo; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Ombrabulin (AVE8062) — Pharmaceutical form:solution
  Route of administration: intravenous
  Arms: Arm A
Drug: Placebo — Pharmaceutical form:solution
  Route of administration: intravenous
  Arms: Arm B
Drug: Paclitaxel — Pharmaceutical form:solution
  Route of administration: intravenous
Drug: Carboplatin — Pharmaceutical form:solution
  Route of administration: intravenous

SUMMARY:
Primary Objective:

- To demonstrate an improvement in Progression-Free Survival (PFS) for Ombrabulin versus placebo in patients with platinum-sensitive recurrent ovarian cancer (OC) treated with paclitaxel and carboplatin.

Secondary Objectives:

* To compare the overall survival (OS) between the 2 treatment arms
* To compare the objective response rate (RR) between the 2 treatment arms

DETAILED DESCRIPTION:
Treatment will continue until disease progression or unacceptable toxicity or consent withdrawal. A minimum of 6 cycles of the combined therapies should be administered, unless progression occurs before or safety reasons cause the discontinuation of one or two drugs of the combination therapies. In case of no progression, it will be investigator's decision to continue or not the study treatment after 6 cycles according to his clinical practice.

ELIGIBILITY:
Inclusion criteria:

1. Signed informed consent.
2. At least 18 years of age.
3. Histological and/or cytological diagnosis of epithelial ovarian carcinoma, fallopian tube cancer, or primary peritoneal carcinoma.
4. Completion of maximum one previous line of chemotherapy containing a platinum agent. Neoadjuvant/adjuvant treatment that include a surgical procedure will be considered as one line if platinum-based.
5. Documented sensitivity to a platinum based chemotherapy regimen. "Platinum-sensitivity" is defined by a relapse more than 6 months after last dose of platinum-based chemotherapy.
6. Measurable progressive disease: Measurable disease (as defined by RECIST 1.1) is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be at least 10mm when measured by computed tomography (CT) or magnetic resonance imaging (MRI). Lymph nodes must be >15 mm in short axis when measured by CT or MRI. In case of a single measurable lesion, this should not be previously irradiated.
7. ECOG performance status ≤2
8. Life expectancy more than 12 weeks

Exclusion criteria:

1. History of uncontrolled brain metastases, spinal cord compression, or carcinomatous meningitis.
2. History of another neoplasm. Adequately treated basal cell or squamous skin cancer, or in situ cervical cancer, or any other cancer from which the patient has been disease-free for >5 years are allowed.
3. Participation in another clinical trial and any concurrent treatment with any investigational drug or anti-tumor therapy or radiotherapy within 21 days prior to randomization (or 28 days for those therapies with a schedule of administration every 4 weeks and except for nitrosoureas, mitomycin which may not be used up to 6 weeks prior to the first cycle provided that patients do not have residual signs of any toxicity). No wash-out is required for hormonotherapy which has to be discontinued before the first cycle.
4. Any severe acute or chronic medical condition, which could impair the ability of the patient to participate in the study or interfere with interpretation of study results.
5. Pregnancy or breast-feeding. Positive serum or urine pregnancy test prior to randomization.
6. Patient with reproductive potential who do not agree to use accepted and effective method of contraception during the study treatment period and for at least 6 months after the completion of the study treatment. The definition of "effective method of contraception" will be based on the investigator's judgment. Effective method of contraception should also be adapted to local regulations.
7. Inadequate organ function including: neutrophils <1.5 x 10^9/L; platelets <100 x 10^9/L; creatinine ≥ 1.5 ULN. If creatinine ≥ ULN, the calculated creatinine clearance should be ≥ 60 ml/min (as per Cockcroft Formula). Total bilirubin not within normal limit and ALT/AST/AP >2.5 times the upper normal limits of the institutional norms. An increase of AP up to grade 2 would be accepted only if this increase is related to the presence of bone metastases. Bone specific isoenzyme AP should be evaluated.
8. Urine protein-creatinin ratio (UPCR) >1 (urinanalysis on morning spot urine) or proteinuria >500 mg/24h
9. Pre-existing peripheral neuropathy > grade 1 according to the NCI CTCAE V.4.03
10. Pre-existing hearing impairment > grade 1
11. Known hypersensitivity due to taxanes and /or polysorbate 80 or any other compound/excipients of the study drug combination
12. Discontinuation of previous treatment with paclitaxel and/or carboplatin for toxicity reason
13. Other serious illness or medical conditions such as (but not restricted):

    * Active infection
    * Superior vena cava syndrome
    * Pericardial effusion requiring intervention (drainage)
14. Documented medical history of myocardial infarction, documented angina pectoris, arrhythmia especially severe conduction disorder such as second or third-degree atrioventricular block, stroke, or history of arterial or venous thrombo-embolism within the past 6 months still requiring anticoagulants.
15. Cardiac Troponin at levels that exceed the normal ranges values defined by the laboratory
16. Uncontrolled hypertension within 3 months prior to study treatment or patient with organ damage related to hypertension.
17. Patient with LVEF value lower than institution inferior normal limit, evaluated by echocardiography or angiocardiography
18. 12-lead ECG:

    * Infarction Q-wave,
    * ST segment depression or elevation ≥1 mm in at least 2 contiguous leads
    * QT/QTc-Time > 450ms

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2011-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | approximately 24 months

SECONDARY OUTCOMES:
Overall Survival (OS) | approximately 24 months
Objective Response Rate (RR) | approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (38):
- United States (5):
  - Investigational Site Number 840007, Burbank, California
  - Investigational Site Number 840001, New Haven, Connecticut
  - Investigational Site Number 840202, Fort Meyers, Florida
  - Investigational Site Number 840009, Atlanta, Georgia
  - Investigational Site Number 840002, Boston, Massachusetts
- Belgium (4):
  - Investigational Site Number 056002, Haine-Saint-Paul
  - Investigational Site Number 056005, Kortrijk
  - Investigational Site Number 056001, Leuven
  - Investigational Site Number 056003, Namur
- Czechia (4):
  - Investigational Site Number 203003, Nový Jičín
  - Investigational Site Number 203002, Olomouc
  - Investigational Site Number 203001, Prague
  - Investigational Site Number 203004, Zlín
- France (5):
  - Investigational Site Number 250006, Bordeaux
  - Investigational Site Number 250004, Caen
  - Investigational Site Number 250001, Lyon
  - Investigational Site Number 250002, Paris
  - Investigational Site Number 250003, Villejuif
- Investigational Site Number 276001, München, Germany
- Italy (3):
  - Investigational Site Number 380004, Genova
  - Investigational Site Number 380003, Milan
  - Investigational Site Number 380001, Roma
- Poland (5):
  - Investigational Site Number 616002, Krakow
  - Investigational Site Number 616004, Poznan
  - Investigational Site Number 616003, Rybnik
  - Investigational Site Number 616005, Warsaw
  - Investigational Site Number 616001, Warsaw
- Russia (4):
  - Investigational Site Number 643002, Moscow
  - Investigational Site Number 643003, Moscow
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643004, Saint Petersburg
- Spain (3):
  - Investigational Site Number 724002, Barcelona
  - Investigational Site Number 724003, Madrid
  - Investigational Site Number 724001, Madrid
- Ukraine (4):
  - Investigational Site Number 804003, Dnipropetrovsk
  - Investigational Site Number 804005, Donetsk
  - Investigational Site Number 804004, Kharkiv
  - Investigational Site Number 804002, Lviv